CLINICAL TRIAL: NCT00402103
Title: A 54-week, Open-label, Multicenter Study to Assess the Long-term Safety and Tolerability of the Combination of Aliskiren 300 mg / Amlodipine 10 mg in Patients With Essential Hypertension
Brief Title: An Assessment of Long Term Safety of the Combination of Aliskiren / Amlodipine in Patients With High Blood Pressure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPA100A2301
Record Dates: First submitted 2006-11-18; First posted 2006-11-22 (Estimated); Results first posted 2011-01-11 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Hypertension
Keywords: Hypertension, aliskiren, amlodipine, HCTZ, blood pressure
MeSH Terms: conditions — Hypertension | interventions — aliskiren; Amlodipine; Hydrochlorothiazide

ARMS (2):
- Aliskiren/Amlodipine (Experimental)
  Interventions: Drug: Aliskiren; Drug: Amlodipine
- Aliskiren/Amlodipine/HCTZ (Experimental)
  Interventions: Drug: Aliskiren; Drug: Amlodipine; Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Aliskiren — All patients received aliskiren 150 mg for the first two weeks; dose was then force-titrated to aliskiren 300 mg for 52 weeks duration
Drug: Amlodipine — All patients received amlodipine 5 mg for the first two weeks; dose was then force-titrated to amlodipine 10 mg for 52 weeks duration
Drug: Hydrochlorothiazide — Optional addition of Hydrochlorothiazide (HCTZ)of 12.5 mg with increase to 25 mg was allowed for patients not adequately controlled.
  Arms: Aliskiren/Amlodipine/HCTZ

SUMMARY:
To assess the long-term (6 month and 12 month) safety of the combination of aliskiren 300 mg / amlodipine 10 mg in patients with essential hypertension (Mean Sitting Diastolic Blood Pressure [msDBP] ≥ 90 mmHg and < 110 mmHg).

ELIGIBILITY:
Inclusion Criteria:

* Outpatients 18 years of age or older
* Male or female patients are eligible
* For newly diagnosed/untreated patients with essential hypertension defined as msDBP ≥ 90 and < 110 mmHg at Visit 1 and Visit 4
* For previously treated patients with essential hypertension defined as msDBP ≥ 90 and < 110 mmHg after 2 to 4 weeks of washout (Visit 4)

Exclusion Criteria:

* Severe hypertension
* History or evidence of a secondary form of hypertension
* History of Hypertensive encephalopathy or cerebrovascular accident.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Actual)
Dates: Start 2006-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis
Locations (8):
- Investigative Site, Santa Fe, New Mexico, United States
- Investigator Site, Investigative Site, Belgium
- Investigative Center, Investigative Center, Denmark
- Investigative Site, Investigative Site, Finland
- Investigative Center, Investigative Center, Germany
- Investigative Site, Investigative Site, Iceland
- Investigative Site, Investigative Site, India
- Investigative Site, Investigative Site, Switzerland

REFERENCES:
- [Derived] Littlejohn TW 3rd, Trenkwalder P, Hollanders G, Zhao Y, Liao W. Long-term safety, tolerability and efficacy of combination therapy with aliskiren and amlodipine in patients with hypertension. Curr Med Res Opin. 2009 Apr;25(4):951-9. doi: 10.1185/03007990902785845. PMID 19257800

RESULTS

PARTICIPANT FLOW:
Groups:
- Aliskiren/Amlodipine: Aliskiren and Amlodipine tablets once a day in the morning
- Aliskiren/Amlodipine/HCTZ: Aliskiren and Amlodipine tablets and HCTZ capsules once a day in the morning
Period: Overall Study
Arm/Group | Aliskiren/Amlodipine | Aliskiren/Amlodipine/HCTZ
Started | 470 | 86
Completed | 379 | 73
Not Completed | 91 | 13
Not completed — Adverse Event | 60 | 7
Not completed — Unsatisfactory therapeutic effect | 1 | 2
Not completed — Condition no longer requires study drug | 2 | 0
Not completed — Protocol Deviation | 8 | 0
Not completed — Patient withdrew consent | 12 | 1
Not completed — Lost to Follow-up | 6 | 3
Not completed — Administrative problems | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren/Amlodipine | Aliskiren/Amlodipine/HCTZ | Total
Number analyzed (Participants) | 470 | 86 | 556
Age Continuous [Mean (Standard Deviation); unit: years] | 54.2 (11.66) | 55.7 (11.33) | 54.4 (11.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196 | 30 | 226
  Male | 274 | 56 | 330

OUTCOME MEASURES:

1. Primary Outcome: Overall Percentage of Patients With Adverse Events
Time Frame: 52 weeks
Population: Treated Population
Measure: Number; unit: Percentage of Participants
Groups:
- Aliskiren 150mg/ Amlodipine 5mg Alone: Aliskiren 150mg and Amlodipine 5mg tablets once a day in the morning
- Aliskiren 300mg/ Amlodipine 10mg Alone: Aliskiren 300mg and Amlodipine 10mg tablets once a day in the morning
- Aliskiren 300mg/ Amlodipine 10mg/ HCTZ: Aliskiren 300mg and Amlodipine 10mg tablets and HCTZ capsules once a day in the morning
Arm/Group | Aliskiren 150mg/ Amlodipine 5mg Alone | Aliskiren 300mg/ Amlodipine 10mg Alone | Aliskiren 300mg/ Amlodipine 10mg/ HCTZ
Number analyzed (Participants) | 556 | 546 | 86
Percentage of Participants | 23.6 | 71.2 | 57.0

2. Secondary Outcome: Change in Mean Sitting Diastolic Blood Pressure (msDBP)From Baseline to the Indicated Time Points
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 10, Week 14, Week 28, Week 41 and Week 54
Population: Treated population, Last observation carried forward (LOCF). Total combined treated patients are 556 out of which 470 patients are treated with Aliskiren and Amlodipine combination only and 86 patients are treated with Ali/Amlo/HCTZ combination.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Aliskiren/Amlodipine | Aliskiren/Amlodipine/HCTZ
Number analyzed (Participants) | 470 | 86
mm Hg
  Week 2 (Visit 5) | -8.7 (6.94) | -5.9 (6.05)
  Week 4 (Visit 6) | -14.0 (6.88) | -11.9 (5.58)
  Week 6 (Visit 7) | -15.7 (6.96) | -11.5 (7.36)
  Week 10 (Visit 8) | -16.3 (6.69) | -9.3 (7.22)
  Week 14 (Visit 9) | -17.1 (6.84) | -13.1 (7.64)
  Week 28 (Visit 10) | -16.7 (7.15) | -14.7 (8.22)
  Week 41 (Visit 11) | -17.0 (7.26) | -15.4 (6.86)
  Week 54 (Visit 12) | -16.3 (7.13) | -15.3 (6.55)
  Week 54 (Visit 12) (LOCF) | -15.7 (7.61) | -14.2 (7.90)

3. Secondary Outcome: Percentage of Patients Achieving a Blood Pressure Control Target of <140/90 mmHg
Time Frame: Baseline, Week 2, Week 10, Week 28 and Week 54
Population: as for outcome 2
Measure: Number; unit: Percentage of patients
Arm/Group | Aliskiren/Amlodipine | Aliskiren/Amlodipine/HCTZ
Number analyzed (Participants) | 470 | 86
Percentage of patients
  Week 2 (Visit 5) | 35.3 (88.0) | 8.1
  Week 10 (Visit 8) | 88.0 | 16.3
  Week 28 (Visit 10) | 88.2 | 56.8
  Week 54 (Visit 12) | 82.0 | 62.2
  Week 54 (Visit 12) (LOCF) | 77.3 | 58.1

4. Secondary Outcome: Percentage of Patients Achieving a Response in Mean Sitting Diastolic Blood Pressure (msDBP)
Time Frame: Baseline, Week 2, Week 10, Week 28 and Week 54
Population: as for outcome 2
Measure: Number; unit: Percentage of patients
Arm/Group | Aliskiren/Amlodipine | Aliskiren/Amlodipine/HCTZ
Number analyzed (Participants) | 470 | 86
Percentage of patients
  Week 2 (Visit 5) | 61.2 | 38.4
  Week 10 (Visit 8) | 96.8 | 61.6
  Week 28 (Visit 10) | 95.9 | 85.2
  Week 54 (Visit 12) | 93.2 | 89.2
  Week 54 (Visit 12) (LOCF) | 90.6 | 84.9

ADVERSE EVENTS:
Arm/Group | Aliskiren 150mg/ Amlodipine 5mg Alone | Aliskiren 300mg/ Amlodipine 10mg Alone | Aliskiren 300mg/ Amlodipine 10mg/ HCTZ
Serious Adverse Events (participants affected / at risk) | 0/556 | 13/546 | 2/86
Other Adverse Events (participants affected / at risk) | 14/556 | 138/546 | 21/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren 150mg/ Amlodipine 5mg Alone (N=556) | Aliskiren 300mg/ Amlodipine 10mg Alone (N=546) | Aliskiren 300mg/ Amlodipine 10mg/ HCTZ (N=86)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0
Amoebiasis (Infections and infestations) | 0 | 1 | 0
Gangrene (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pubic rami fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren 150mg/ Amlodipine 5mg Alone (N=556) | Aliskiren 300mg/ Amlodipine 10mg Alone (N=546) | Aliskiren 300mg/ Amlodipine 10mg/ HCTZ (N=86)
Oedema peripheral (General disorders) | 8 | 108 | 12
Upper respiratory tract infection (Infections and infestations) | 5 | 32 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.